CLINICAL TRIAL: NCT02803307
Title: A Randomized, Open-label, Parallel, Phase I/II Single-Dose Administration Trial of TLC599 in Subjects With Osteoarthritis of the Knee
Brief Title: Single-Dose Administration Trial of TLC599 in Osteoarthritis of the Knee
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Taiwan Liposome Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TLC599A1001
Record Dates: First submitted 2016-05-23; First posted 2016-06-16 (Estimated); Results first posted 2022-05-06 (Actual); Last update posted 2022-05-06 (Actual); Status verified 2022-05

CONDITIONS: Osteoarthritis of the Knee
Keywords: osteoarthritis of the knee; TLC599; Dexamethasone; DSP
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 6 mg TLC599 (Experimental): 6 mg DSP with 50 μmol PL
  Interventions: Drug: TLC599
- 12 mg TLC599 (Experimental): 12 mg DSP with 100 μmol PL
  Interventions: Drug: TLC599

INTERVENTIONS:
Drug: TLC599 — Single dose via intra-articular injection

SUMMARY:
This trial is a multi-site, randomized, open-label, parallel, and single-dose administration study to investigate the safety and efficacy of TLC599 in subjects with osteoarthritis of the knee.

DETAILED DESCRIPTION:
Protocol No: TLC599A1001

Name of Finished Product: TLC599

Title of Study:

A Randomized, Open-label, Parallel, Phase I/II Single-Dose Administration trial of TLC599 in Subjects with Osteoarthritis (OA) of the Knee

Methodology This trial is a multi-site, randomized, open-label, parallel, and single-dose administration study to investigate the safety and efficacy of TLC599 in subjects with osteoarthritis of the knee.

Study duration:

The trial will last 14 weeks including a 14-day screening period and a 12-week follow-up period.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female subjects, at least 20 years of age
2. Documented diagnosis of OA of the knee for at least 6 months
3. At least a grade 2 severity based on the Kellgren and Lawrence Grading Scale
4. VAS score of ≥ 4 at baseline

Exclusion Criteria:

1. Subjects who received systemic corticosteroids for the last 30 days prior to baseline
2. Subjects who received non-steroidal anti-inflammatory drug (NSAID), analgesics, or rehabilitations therapy within 7 days prior to baseline
3. History of rheumatoid arthritis or other autoimmune disease
4. Clinical signs and symptoms of acute infection or infection related inflammation in the other knee before dosing
5. History of infective arthritis, suspected or concurrent infection, or suspected or confirmed crystal diseases (gout or pseudogout) of the study knee
6. Concurrent systemic active or uncontrolled infectious disease
7. A history of treated malignancy which is disease free for ≤ 5 years. (The malignancy does not include non-basal-cell carcinoma of skin or carcinoma-insitu of the uterine cervix)
8. History of acquired or congenital immunodeficiency diseases
9. Platelet count < 80,000/μl, or blood coagulation disorders, including subjects with hemophilia, decompensated liver cirrhosis or uremia
10. Stroke or myocardial infarction within 3 months prior to the screening visit
11. Use of intra-articular corticosteroid, hyaluronic acid, or other intra-articular injection in the study knee joint within 3 months prior to the screening visit
12. Unstable study knee joint, including anterior cruciate ligament, any surgery to the study knee within the 12 months prior to the screening visit, and any prior arthroscopic or open surgery of the study knee or any planned/anticipated surgery during the study period
13. Any skin lesion/breakdown at the anticipated injection site or any condition that impairs penetration of the study knee joint space
14. Female subjects who are pregnant, nursing, planning pregnancy, or who are of childbearing potential and not using reliable means of contraception 15.Known allergy or hypersensitivity to the study drug or its components

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2015-06 (Actual); Primary Completion 2016-11 (Actual); Study Completion 2016-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Carl Brown, PhD, Study Director — Taiwan Liposome Company
Locations (3):
- Taiwan (3):
  - MacKay Memorial Hospital, Taipei
  - Taipei Medical University Hospital, Taipei
  - Taipei Veterans General Hospital, Taipei

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | 6 mg TLC599 | 12 mg TLC599
Started | 20 | 20
Completed | 20 | 20
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 6 mg TLC599 | 12 mg TLC599 | Total
Number analyzed (Participants) | 20 | 20 | 40
Age, Continuous [Mean (Standard Deviation); unit: years] | 66.70 (10.04) | 68.10 (8.03) | 67.40 (9.00)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18 | 14 | 32
  Male | 2 | 6 | 8
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 20 | 20 | 40
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Taiwan | 20 | 20 | 40
Kellgren-Lawrence grade [Count of Participants; unit: Participants] — The Kellgren-Lawrence (K-L) grading system is a method of classifying the severity of knee osteoarthritis (OA) using 5 grades:
  Grade 0: No radiographic features of OA are present; Grade 1: Doubtful joint space narrowing (JSN) and possible osteophytic lipping; Grade 2: Definite osteophytes and possible JSN on posteroanterior weight-bearing radiograph; Grade 3: Multiple osteophytes, definite JSN, sclerosis, possible bony deformity; Grade 4: Large osteophytes, marked JSN, severe sclerosis and definite bony deformity.
  Participants
    Grade 0 | 0 | 0 | 0
    Grade 1 | 0 | 0 | 0
    Grade 2 | 7 | 5 | 12
    Grade 3 | 10 | 10 | 20
    Grade 4 | 3 | 5 | 8

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment-Emergent Adverse Events (TEAEs)
Description: Number of participants with at least one TEAE
Time Frame: up to 12 weeks after dosing
Measure: Count of Participants; unit: Participants
Arm/Group | 6 mg TLC599 | 12 mg TLC599
Number analyzed (Participants) | 20 | 20
Participants | 9 | 9

ADVERSE EVENTS:
Time Frame: 12 weeks
Arm/Group | 6 mg TLC599 | 12 mg TLC599
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/20
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/20
Other Adverse Events (participants affected / at risk) | 9/20 | 9/20
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | 6 mg TLC599 (N=20) | 12 mg TLC599 (N=20)
Angina pectoris (Cardiac disorders) | 0 | 1
Arrhythmia (Cardiac disorders) | 1 | 0
Vertigo (Ear and labyrinth disorders) | 0 | 1
Abdominal pain upper (Gastrointestinal disorders) | 0 | 1
Colitis (Gastrointestinal disorders) | 0 | 1
Gastric disorder (Gastrointestinal disorders) | 0 | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 1
Pyrexia (General disorders) | 1 | 0
Cholelithiasis (Hepatobiliary disorders) | 0 | 1
Bronchitis (Infections and infestations) | 0 | 1
Influenza (Infections and infestations) | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 1 | 0
Urinary tract infection (Infections and infestations) | 1 | 0
Vaginal infection (Infections and infestations) | 0 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 3
Hyperlipidaemia (Metabolism and nutrition disorders) | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1
Synovial cyst (Musculoskeletal and connective tissue disorders) | 0 | 1
Dizziness (Nervous system disorders) | 1 | 1
Headache (Nervous system disorders) | 0 | 1
Bronchitis chronic (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Dermatitis contact (Skin and subcutaneous tissue disorders) | 1 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 0
Hypertension (Vascular disorders) | 1 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No